CLINICAL TRIAL: NCT00428597
Title: A Phase III Randomized, Double-Blind Study Of Sunitinib (SU011248, SUTENT) Versus Placebo In Patients With Progressive Advanced/Metastatic Well-Differentiated Pancreatic Islet Cell Tumors
Brief Title: A Study Of Sunitinib Compared To Placebo For Patients With Advanced Pancreatic Islet Cell Tumors
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Refer to Detailed Description.
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer Inc
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A6181111
Record Dates: First submitted 2007-01-29; First posted 2007-01-30 (Estimated); Results first posted 2010-10-11 (Estimated); Last update posted 2010-10-11 (Estimated); Status verified 2010-09

CONDITIONS: Carcinoma, Islet Cell; Carcinoma, Pancreas
MeSH Terms: conditions — Carcinoma, Islet Cell; Pancreatic Neoplasms | interventions — Sunitinib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental)
  Interventions: Drug: sunitinib malate
- B (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: sunitinib malate — * sunitinib malate oral starting dose 37.5 mg daily (continuous dosing).
  * Dose may be decreased to 25 mg daily in case of adverse events.
  * It may be increased to 50 mg daily if no response is seen after 8 weeks on treatment.
  * Dosing to continue until unacceptable toxicity, progression of disease, death, or study termination.
  Arms: A
Drug: Placebo — Placebo to match sunitinib taken daily (oral) on the same schedule as active agent below.
  Arms: B

SUMMARY:
This study randomized patients with advanced pancreatic islet cell tumors to receive either sunitinib or placebo. Patients who were randomized to sunitinib received 37.5 mg of sunitinib daily, those randomized to placebo received a tablet that looked similar but had no active drug. Neither the patient or the doctor knew whether the patient was receiving sunitinib or placebo. Patients were followed to determine the status and size of their tumors, survival, quality of life and safety of the drug.

The study was designed to detect a 50% improvement in median PFS[Progression Free Survival] with 90% power and was to enroll 340 subjects. An interim analysis was planned when 130 events had occurred, and the final analysis was to be conducted when 260 events had occurred.

Study A6181111 was stopped early during the enrollment period because of a clear and clinically meaningful improvement in efficacy for the sunitinib treatment arm as recommended by the DMC [Data Monitoring Committee]. The actual number of subjects enrolled was 171 and the actual number of PFS events recorded was 81 PFS events. The decision to terminate the study was not based on safety concerns related to sunitinib administration.

DETAILED DESCRIPTION:
The study was terminated on 11 March 2009 because the independent Data Monitoring Committee determined that the study had met its primary endpoint in demonstrating improvement in progression-free survival. The decision to terminate the trial was not based on safety concerns related to sunitinib administration.

ELIGIBILITY:
Inclusion Criteria:

* Well-differentiated advanced/metastatic pancreatic islet cell tumor
* Tumor has shown progression within the past year.

Exclusion Criteria:

* Current treatment with any chemotherapy, chemoembolization therapy, immunotherapy, or investigational anticancer agent other than somatostatin analogues
* Prior treatment with any tyrosine kinase inhibitors or anti-VEGF[Vascular endothelial growth factor] angiogenic inhibitors.
* Prior treatment with non-VEGF-targeted angiogenic inhibitors is permitted

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 171 (Actual)
Dates: Start 2007-06; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (40):
- United States (9):
  - Pfizer Investigational Site, Aurora, Colorado
  - Pfizer Investigational Site, Iowa City, Iowa
  - Pfizer Investigational Site, Worcester, Massachusetts
  - Pfizer Investigational Site, City of Saint Peters, Missouri
  - Pfizer Investigational Site, Creve Coeur, Missouri
  - Pfizer Investigational Site, St Louis, Missouri
  - Pfizer Investigational Site, Austin, Texas
  - Pfizer Investigational Site, Georgetown, Texas
  - Pfizer Investigational Site, Norfolk, Virginia
- Pfizer Investigational Site, Perth, Western Australia, Australia
- Belgium (2):
  - Pfizer Investigational Site, Brussels
  - Pfizer Investigational Site, Leuven
- Canada (4):
  - Pfizer Investigational Site, Vancouver, British Columbia
  - Pfizer Investigational Site, Halifax, Nova Scotia
  - Pfizer Investigational Site, Toronto, Ontario
  - Pfizer Investigational Site, Montreal, Quebec
- France (7):
  - Pfizer Investigational Site, Paris, Be1 05677
  - Pfizer Investigational Site, Paris, Cedex
  - Pfizer Investigational Site, Clichy, France
  - Pfizer Investigational Site, Bordeaux
  - Pfizer Investigational Site, Lyon
  - Pfizer Investigational Site, Marseille
  - Pfizer Investigational Site, Rennes
- Germany (6):
  - Pfizer Investigational Site, Bad Berka
  - Pfizer Investigational Site, Berlin
  - Pfizer Investigational Site, Heidelberg
  - Pfizer Investigational Site, Lübeck
  - Pfizer Investigational Site, Marburg
  - Pfizer Investigational Site, Ulm
- Italy (3):
  - Pfizer Investigational Site, Cremona
  - Pfizer Investigational Site, Milan
  - Pfizer Investigational Site, Rozzano (MI)
- Pfizer Investigational Site, Seoul, South Korea
- Spain (2):
  - Pfizer Investigational Site, Barcelona, Barcelona
  - Pfizer Investigational Site, Madrid, Madrid
- Taiwan (2):
  - Pfizer Investigational Site, Kwei-Shan, Taoyuan
  - Pfizer Investigational Site, Taipei
- United Kingdom (3):
  - Pfizer Investigational Site, Leeds
  - Pfizer Investigational Site, Liverpool
  - Pfizer Investigational Site, Manchester

REFERENCES:
- [Derived] Fazio N, Kulke M, Rosbrook B, Fernandez K, Raymond E. Updated Efficacy and Safety Outcomes for Patients with Well-Differentiated Pancreatic Neuroendocrine Tumors Treated with Sunitinib. Target Oncol. 2021 Jan;16(1):27-35. doi: 10.1007/s11523-020-00784-0. Epub 2021 Jan 7. PMID 33411058
- [Derived] Lamarca A, Barriuso J, Kulke M, Borbath I, Lenz HJ, Raoul JL, Meropol NJ, Lombard-Bohas C, Posey J, Faivre S, Raymond E, Valle JW. Determination of an optimal response cut-off able to predict progression-free survival in patients with well-differentiated advanced pancreatic neuroendocrine tumours treated with sunitinib: an alternative to the current RECIST-defined response. Br J Cancer. 2018 Jan;118(2):181-188. doi: 10.1038/bjc.2017.402. Epub 2017 Nov 21. PMID 29161241
- [Derived] Vinik A, Bottomley A, Korytowsky B, Bang YJ, Raoul JL, Valle JW, Metrakos P, Horsch D, Mundayat R, Reisman A, Wang Z, Chao RC, Raymond E. Patient-Reported Outcomes and Quality of Life with Sunitinib Versus Placebo for Pancreatic Neuroendocrine Tumors: Results From an International Phase III Trial. Target Oncol. 2016 Dec;11(6):815-824. doi: 10.1007/s11523-016-0462-5. PMID 27924459
- [Derived] Faivre S, Niccoli P, Castellano D, Valle JW, Hammel P, Raoul JL, Vinik A, Van Cutsem E, Bang YJ, Lee SH, Borbath I, Lombard-Bohas C, Metrakos P, Smith D, Chen JS, Ruszniewski P, Seitz JF, Patyna S, Lu DR, Ishak KJ, Raymond E. Sunitinib in pancreatic neuroendocrine tumors: updated progression-free survival and final overall survival from a phase III randomized study. Ann Oncol. 2017 Feb 1;28(2):339-343. doi: 10.1093/annonc/mdw561. PMID 27836885
- [Derived] Raymond E, Dahan L, Raoul JL, Bang YJ, Borbath I, Lombard-Bohas C, Valle J, Metrakos P, Smith D, Vinik A, Chen JS, Horsch D, Hammel P, Wiedenmann B, Van Cutsem E, Patyna S, Lu DR, Blanckmeister C, Chao R, Ruszniewski P. Sunitinib malate for the treatment of pancreatic neuroendocrine tumors. N Engl J Med. 2011 Feb 10;364(6):501-13. doi: 10.1056/NEJMoa1003825. PMID 21306237
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A6181111&StudyName=A%20Study%20Of%20Sunitinib%20Compared%20To%20Placebo%20For%20Patients%20With%20Advanced%20Pancreatic%20Islet%20Cell%20Tumors

RESULTS

PARTICIPANT FLOW:
Groups:
- Sunitinib: Oral sunitinib 37.5 milligrams (mg) once daily on a continuous daily dosing schedule.
- Placebo: Matching placebo.
Period: Overall Study
Arm/Group | Sunitinib | Placebo
Started | 86 | 85
Received Treatment | 83 | 82
Completed | 0 | 0
Not Completed | 86 | 85
Not completed — Randomized but not treated | 3 | 3
Not completed — Objective Progression or Relapse | 19 | 47
Not completed — Study Terminated by Sponsor | 41 | 16
Not completed — Adverse Event | 15 | 7
Not completed — Global Deterioration of Health Status | 1 | 5
Not completed — Protocol Violation | 2 | 1
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Other | 1 | 1
Not completed — Lost to Follow-up | 0 | 1
Not completed — Pregnancy | 1 | 0
Not completed — Death | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Sunitinib: Oral sunitinib 37.5 mg once daily on a continuous daily dosing schedule.
- Total: Total of all reporting groups
Arm/Group | Sunitinib | Placebo | Total
Number analyzed (Participants) | 86 | 85 | 171
Age, Customized [Number; unit: participants]
  Between 18 and 44 years | 19 | 17 | 36
  Between 45 and 64 | 45 | 45 | 90
  >=65 years | 22 | 23 | 45
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44 | 45 | 89
  Male | 42 | 40 | 82

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS)
Description: Time from randomization to first progression of disease (PD) or death for any reason in the absence of documented PD. PFS was calculated as (first event date minus first randomization date +1) divided by 30.4.
Time Frame: From time of randomization through Day 1 of Week 5, Week 9, and then every 8 weeks thereafter until disease progression or death
Population: Intent-to-treat (ITT) population = all subjects who were randomized.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Sunitinib | Placebo
Number analyzed (Participants) | 86 | 85
Months | 11.4 [7.4 to 19.8] | 5.5 [3.6 to 7.4]
Statistical Analysis 1: Comparison: Sunitinib vs Placebo; Test type: Superiority or Other; p = 0.000118, Log Rank — Log-rank test statistic and 2-sided p-value from the unstratified log-rank test; Hazard Ratio (HR) = 0.418, 95% CI 2-sided [0.263 to 0.662] — Hazard ratio based on the Cox Proportional hazards model

2. Secondary Outcome: Number of Subjects With Objective Response
Description: Objective response = subjects with confirmed complete response (CR) or partial response (PR) according to Response Evaluation Criteria in Solid Tumors (RECIST) for at least 4 weeks, confirmed by repeat tumor assessments. A CR was defined as the disappearance of all target lesions. A PR was defined as a > = 30% decrease in the sum of the longest dimensions of the target lesions taking as a reference the baseline sum longest dimensions.
Time Frame: From time of randomization through Day 1 of Week 5, 9, and every 8 weeks thereafter
Population: ITT. No placebo subjects had objective response.
Measure: Number; unit: participants
Arm/Group | Sunitinib
Number analyzed (Participants) | 86
participants | 8
Statistical Analysis 1: Comparison: Sunitinib; Test type: Superiority or Other; Objective Response Rate (ORR) (percent) = 9.3, 95% CI 2-sided [4.1 to 17.5] — Confidence interval (CI) using exact method based on binomial distribution

3. Secondary Outcome: Duration of Response (DR)
Description: Time in months from the first documentation of objective tumor response to objective tumor progression or death due to any cause. DR was calculated as (the date of the first documentation of objective tumor progression or death due to any cause minus the date of the first CR or PR that was subsequently confirmed plus 1) divided by 30.4.
Time Frame: From start of treatment through Day 1 of Week 5, 9, and every 8 weeks thereafter until disease progression or death due to any cause
Population: ITT. DR was calculated for the subgroup of subjects with objective response. 8 sunitinib subjects reported CR or PR response and were analyzed for DR; no placebo subjects reported CR or PR.
Measure: Median (Full Range); unit: Months
Arm/Group | Sunitinib
Number analyzed (Participants) | 8
Months | 8.1 [1.0 to 15.0]

4. Secondary Outcome: Time-to-Tumor Response (TTR)
Description: Time from randomization to the first documentation of objective tumor response (CR or PR) that was subsequently confirmed.
Time Frame: From time of randomization through Day 1 of Week 5, 9, and every 8 weeks thereafter
Population: ITT. TTR was calculated for the subgroup of subjects with objective response. 8 sunitinib subjects reported CR or PR response and were analyzed for TTR; no placebo subjects reported CR or PR.
Measure: Median (Full Range); unit: Months
Arm/Group | Sunitinib
Number analyzed (Participants) | 8
Months | 3.1 [0.8 to 11.1]

5. Secondary Outcome: Overall Survival (OS)
Description: Time in months from time of randomization to date of death due to any cause. The median number of months is provided; however, the study was terminated early. OS data was not mature by the time of analysis. Median OS time cannot be accurately estimated by Kaplan-Meier method for either treatment arm.
Time Frame: From start of study treatment up to 22 months
Population: ITT. The median OS in months could not be calculated for placebo.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Sunitinib
Number analyzed (Participants) | 86
months | 20.6 [20.6 to NA] — The upper confidence interval was not reached.
Statistical Analysis 1: Comparison: Sunitinib; Test type: Superiority or Other; p = 0.0204, Log Rank — 2-sided p-value from the unstratified log-rank test; Hazard Ratio (HR) = 0.409, 95% CI 2-sided [0.187 to 0.894] — Hazard ratio based on the Cox Proportional hazards model

6. Secondary Outcome: European Organization for Research and Treatment of Cancer Quality of LifeQuestionnaire (EORTC QLQ-C30) - Global Quality of Life (QoL) Subscale
Description: EORTC QLQ-C30 scales: global health/QoL, functional domains (physical, role, cognitive, emotional, social), and symptom scales/items (fatigue, nausea and vomiting, pain, dyspnea, insomnia, appetite loss, constipation, diarrhea). Recall period: past week; response range: not at all to very much, global/QOL range: very poor to excellent. Scale score range: 0 to 100. Higher functional/global QoL score = better functioning and higher symptom score = greater degree of symptoms.
Time Frame: Day 1 and every 4 weeks thereafter (Day 1 of each 4-week cycle) and at end of treatment/withdrawal
Population: Patient Reported Outcome (PRO) population=subjects from the ITT population who had completed at least 1 EORTC QLQ-C30 assessment while on treatment. n=number of subjects with EORTC QLQ-C30 score at each specified time point. Data in cycles beyond Cycle 10 are not reported due to few subjects and lack of statistical reliability.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Sunitinib | Placebo
Number analyzed (Participants) | 73 | 71
scores on a scale
  Cycle 1 (n=66, 66) | 67.0 (20.3) [58.7 to 66.1] | 64.0 (22.7) [57.2 to 65.3]
  Cycle 2 (n=68, 66) | 62.1 (19.9) | 62.6 (23.6)
  Cycle 3 (n=60, 56) | 62.6 (20.7) | 63.5 (25.1)
  Cycle 4 (n=55, 43) | 62.0 (21.8) | 61.6 (23.3)
  Cycle 5 (n=48, 40) | 63.5 (21.9) | 61.7 (25.4)
  Cycle 6 (n=42, 31) | 66.9 (22.0) | 56.7 (29.8)
  Cycle 7 (n=37, 28) | 66.2 (23.0) | 64.6 (23.4)
  Cycle 8 (n=33, 22) | 65.9 (23.6) | 62.1 (23.2)
  Cycle 9 (n=33, 18) | 67.2 (19.1) | 64.4 (22.1)
  Cycle 10 (n=29, 14) | 71.0 (20.1) | 59.5 (24.0)
Statistical Analysis 1: Comparison: Sunitinib vs Placebo; Cycle 2 through Cycle 10; Test type: Superiority or Other; p = 0.6799, Repeated Measures Mixed-Effects Model — From repeated measures mixed-effects with intercept term, treatment, time from first dose, treatment-by-time interaction and baseline score (intercept and time from dose as random effects). No p-value adjustments were made for multiple comparisons; Mean Difference (Final Values) = 1.1543, 95% CI 2-sided [-4.3 to 6.6] — Estimated mean difference with 95% CI and p-value were obtained from the repeated measures mixed-effects model using data from Cycle 2 through Cycle 10

7. Secondary Outcome: EORTC QLQ-C30 - Cognitive Functioning Subscale
Description: as for outcome 6
Time Frame: Day 1 and every 4 weeks thereafter (Day 1 of each 4-week cycle) and at end of treatment/withdrawal
Population: PRO population. n=number of subjects with EORTC QLQ-C30 score at each specified time point. Data in cycles with less than 10 subjects are not reported due to lack of statistical reliability.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Sunitinib | Placebo
Number analyzed (Participants) | 73 | 71
scores on a scale
  Cycle 1 (n=67, 66) | 87.1 (16.6) | 87.1 (18.2)
  Cycle 2 (n=69, 66) | 82.9 (20.0) | 78.5 (24.4)
  Cycle 3 (n=60, 56) | 80.1 (19.9) | 80.8 (22.7)
  Cycle 4 (n=55, 43) | 79.7 (24.2) | 82.6 (18.5)
  Cycle 5 (n=48, 40) | 82.3 (20.2) | 82.9 (21.8)
  Cycle 6 (n=42, 31) | 82.1 (22.5) | 82.3 (20.6)
  Cycle 7 (n=38, 28) | 84.6 (21.0) | 88.1 (15.6)
  Cycle 8 (n=34, 22) | 84.3 (18.3) | 79.5 (23.0)
  Cycle 9 (n=33, 18) | 80.3 (21.8) | 83.3 (18.1)
  Cycle 10 (n=29, 14) | 80.5 (24.0) | 85.7 (19.5)
Statistical Analysis 1: Comparison: Sunitinib vs Placebo; Cycle 2 through Cycle 10; Test type: Superiority or Other; p = 0.6058, Repeated Measures Mixed-Effects Model — [p-value comment as in outcome 6, analysis 1]; Mean Difference (Final Values) = -1.4404, 95% CI 2-sided [-6.9 to 4] — [estimate comment as in outcome 6, analysis 1]

8. Secondary Outcome: EORTC QLQ-C30 - Emotional Functioning Subscale
Description: as for outcome 6
Time Frame: Day 1 and every 4 weeks thereafter (Day 1 of each 4-week cycle) and at end of treatment/withdrawal
Population: PRO population. n=number of subjects with EORTC QLQ-C30 score at each specified time point. Data in cycles beyond Cycle 10 are not reported due to few subjects and lack of statistical reliability.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Sunitinib | Placebo
Number analyzed (Participants) | 73 | 71
scores on a scale
  Cycle 1 (n=67, 66) | 75.2 (23.0) | 73.7 (26.2)
  Cycle 2 (n=69, 66) | 76.2 (22.1) | 73.1 (27.1)
  Cycle 3 (n=60, 56) | 75.3 (20.2) | 70.8 (25.8)
  Cycle 4 (n=55, 43) | 72.2 (23.2) | 76.9 (22.3)
  Cycle 5 (n=48, 40) | 72.6 (25.2) | 75.8 (23.9)
  Cycle 6 (n=42, 31) | 77.8 (23.8) | 72.8 (28.9)
  Cycle 7 (n=38, 28) | 75.3 (28.6) | 80.8 (19.8)
  Cycle 8 (n=34, 22) | 74.0 (30.9) | 76.7 (21.6)
  Cycle 9 (n=33, 18) | 75.4 (23.4) | 75.8 (30.0)
  Cycle 10 (n=29, 14) | 76.4 (23.4) | 76.2 (20.4)
Statistical Analysis 1: Comparison: Sunitinib vs Placebo; Cycle 2 through Cycle 10; Test type: Superiority or Other; p = 0.3008, Repeated Measures Mixed-Effects Model — [p-value comment as in outcome 6, analysis 1]; Mean Difference (Final Values) = -3.5575, 95% CI 2-sided [-10.3 to 3.2] — [estimate comment as in outcome 6, analysis 1]

9. Secondary Outcome: EORTC QLQ-C30 - Physical Functioning Subscale
Description: as for outcome 6
Time Frame: Day 1 and every 4 weeks thereafter (Day 1 of each 4-week cycle) and at end of treatment/withdrawal
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Sunitinib | Placebo
Number analyzed (Participants) | 73 | 71
scores on a scale
  Cycle 1 (n=67, 66) | 83.1 (20.5) | 83.1 (20.6)
  Cycle 2 (n=69, 67) | 77.7 (20.5) | 77.1 (25.9)
  Cycle 3 (n=60, 56) | 78.2 (21.6) | 75.5 (28.5)
  Cycle 4 (n=55, 43) | 77.5 (21.3) | 78.4 (24.5)
  Cycle 5 (n=48, 40) | 78.3 (20.2) | 80.7 (21.9)
  Cycle 6 (n=42, 30) | 80.9 (16.3) | 81.1 (22.3)
  Cycle 7 (n=38, 28) | 80.3 (18.8) | 78.9 (25.4)
  Cycle 8 (n=34, 22) | 79.4 (20.7) | 73.5 (28.1)
  Cycle 9 (n=33, 18) | 78.8 (17.0) | 79.6 (24.8)
  Cycle 10 (n=29, 14) | 81.4 (18.9) | 78.6 (23.3)
Statistical Analysis 1: Comparison: Sunitinib vs Placebo; Cycle 2 through Cycle 10; Test type: Superiority or Other; p = 0.3230, Repeated Measures Mixed-Effects Model — [p-value comment as in outcome 6, analysis 1]; Mean Difference (Final Values) = 2.7911, 95% CI 2-sided [-2.8 to 8.3] — [estimate comment as in outcome 6, analysis 1]

10. Secondary Outcome: EORTC QLQ-C30 - Role Functioning Subscale
Description: as for outcome 6
Time Frame: Day 1 and every 4 weeks thereafter (Day 1 of each 4-week cycle) and at end of treatment/withdrawal
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Sunitinib | Placebo
Number analyzed (Participants) | 73 | 71
scores on a scale
  Cycle 1 (n=67, 66) | 84.3 (23.4) | 77.5 (27.7)
  Cycle 2 (n=69, 67) | 71.6 (28.9) | 68.9 (30.6)
  Cycle 3 (n=60, 56) | 71.0 (26.7) | 70.5 (31.0)
  Cycle 4 (n=55, 43) | 72.1 (28.9) | 73.3 (29.6)
  Cycle 5 (n=48, 41) | 71.5 (27.7) | 75.0 (31.4)
  Cycle 6 (n=42, 31) | 76.6 (26.6) | 66.1 (32.6)
  Cycle 7 (n=38, 28) | 75.7 (28.8) | 72.3 (29.7)
  Cycle 8 (n=34, 22) | 73.0 (29.6) | 66.7 (30.9)
  Cycle 9 (n=33, 18) | 72.2 (24.2) | 67.6 (31.6)
  Cycle 10 (n=29, 14) | 79.9 (22.4) | 70.2 (28.6)
Statistical Analysis 1: Comparison: Sunitinib vs Placebo; Cycle 2 through Cycle 10; Test type: Superiority or Other; p = 0.7113, Repeated Measures Mixed-Effects Model — [p-value comment as in outcome 6, analysis 1]; Mean Difference (Final Values) = 1.5113, 95% CI 2-sided [-6.5 to 9.5] — [estimate comment as in outcome 6, analysis 1]

11. Secondary Outcome: EORTC QLQ-C30 - Social Functioning Subscale
Description: as for outcome 6
Time Frame: Day 1 and every 4 weeks thereafter (Day 1 of each 4-week cycle) and at end of treatment/withdrawal
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Sunitinib | Placebo
Number analyzed (Participants) | 73 | 71
scores on a scale
  Cycle 1 (n=67, 66) | 79.4 (27.2) | 77.0 (31.5)
  Cycle 2 (n=69, 66) | 77.8 (22.1) | 75.0 (31.0)
  Cycle 3 (n=60, 56) | 77.1 (23.1) | 77.2 (28.8)
  Cycle 4 (n=55, 43) | 71.2 (28.4) | 79.8 (26.1)
  Cycle 5 (n=48, 40) | 74.3 (23.8) | 77.3 (30.2)
  Cycle 6 (n=42, 31) | 79.0 (26.3) | 74.7 (31.0)
  Cycle 7 (n=38, 28) | 76.3 (29.2) | 83.9 (25.5)
  Cycle 8 (n=34, 22) | 72.5 (30.4) | 74.2 (31.6)
  Cycle 9 (n=33, 18) | 76.3 (21.7) | 74.1 (33.4)
  Cycle 10 (n=29, 14) | 75.9 (25.8) | 81.0 (24.3)
Statistical Analysis 1: Comparison: Sunitinib vs Placebo; Cycle 2 through Cycle 10; Test type: Superiority or Other; p = 0.6487, Repeated Measures Mixed-Effects Model — [p-value comment as in outcome 6, analysis 1]; Mean Difference (Final Values) = -1.6672, 95% CI 2-sided [-8.9 to 5.5] — [estimate comment as in outcome 6, analysis 1]

12. Secondary Outcome: EORTC QLQ-C30 - Appetite Loss Subscale
Description: as for outcome 6
Time Frame: Day 1 and every 4 weeks thereafter (Day 1 of each 4-week cycle) and at end of treatment/withdrawal
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Sunitinib | Placebo
Number analyzed (Participants) | 73 | 71
scores on a scale
  Cycle 1 (n=67, 66) | 16.9 (25.5) | 18.7 (27.5)
  Cycle 2 (n=69, 67) | 25.1 (33.0) | 20.4 (31.8)
  Cycle 3 (n=60, 56) | 25.0 (34.5) | 23.8 (32.9)
  Cycle 4 (n=55, 43) | 33.3 (34.5) | 22.5 (27.9)
  Cycle 5 (n=48, 41) | 26.4 (33.7) | 24.0 (30.7)
  Cycle 6 (n=42, 31) | 20.6 (30.3) | 23.7 (30.1)
  Cycle 7 (n=38, 28) | 24.6 (29.7) | 19.0 (29.3)
  Cycle 8 (n=34, 21) | 24.5 (31.0) | 30.2 (33.2)
  Cycle 9 (n=33, 18) | 23.2 (27.0) | 22.2 (32.3)
  Cycle 10 (n=29, 14) | 18.4 (29.0) | 21.4 (33.6)
Statistical Analysis 1: Comparison: Sunitinib vs Placebo; Cycle 2 through Cycle 10; Test type: Superiority or Other; p = 0.6545, Repeated Measures Mixed-Effects Model — [p-value comment as in outcome 6, analysis 1]; Mean Difference (Final Values) = 1.8800, 95% CI 2-sided [-6.4 to 10.1] — [estimate comment as in outcome 6, analysis 1]

13. Secondary Outcome: EORTC QLQ-C30 - Constipation Subscale
Description: as for outcome 6
Time Frame: Day 1 and every 4 weeks thereafter (Day 1 of each 4-week cycle) and at end of treatment/withdrawal
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Sunitinib | Placebo
Number analyzed (Participants) | 73 | 71
scores on a scale
  Cycle 1 (n=67, 65) | 14.9 (24.8) | 14.9 (23.6)
  Cycle 2 (n=69, 66) | 8.2 (16.6) | 13.6 (23.4)
  Cycle 3 (n=59, 56) | 9.0 (20.4) | 18.5 (28.4)
  Cycle 4 (n=55, 43) | 9.1 (17.5) | 14.0 (24.4)
  Cycle 5 (n=48, 41) | 7.6 (17.2) | 15.9 (24.7)
  Cycle 6 (n=42, 31) | 11.1 (15.9) | 14.0 (26.9)
  Cycle 7 (n=37, 28) | 9.9 (19.0) | 10.1 (23.7)
  Cycle 8 (n=34, 22) | 11.8 (18.1) | 18.2 (32.1)
  Cycle 9 (n=32, 18) | 10.4 (15.7) | 18.5 (32.8)
  Cycle 10 (n=29, 14) | 13.8 (18.9) | 16.7 (31.4)
Statistical Analysis 1: Comparison: Sunitinib vs Placebo; Cycle 2 through Cycle 10; Test type: Superiority or Other; p = 0.1936, Repeated Measures Mixed-Effects Model — [p-value comment as in outcome 6, analysis 1]; Mean Difference (Final Values) = -4.0035, 95% CI 2-sided [-10 to 2] — [estimate comment as in outcome 6, analysis 1]

14. Secondary Outcome: EORTC QLQ-C30 - Diarrhea Subscale
Description: as for outcome 6
Time Frame: Day 1 and every 4 weeks thereafter (Day 1 of each 4-week cycle) and at end of treatment/withdrawal
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Sunitinib | Placebo
Number analyzed (Participants) | 73 | 71
scores on a scale
  Cycle 1 (n=67, 66) | 20.4 (29.6) | 19.2 (28.1)
  Cycle 2 (n=69, 66) | 37.7 (35.2) | 18.2 (27.5)
  Cycle 3 (n=60, 56) | 34.2 (33.7) | 16.7 (26.2)
  Cycle 4 (n=55, 43) | 38.8 (32.6) | 18.6 (27.5)
  Cycle 5 (n=47, 40) | 42.6 (36.6) | 15.0 (25.0)
  Cycle 6 (n=42, 31) | 38.9 (32.9) | 18.3 (28.3)
  Cycle 7 (n=38, 28) | 41.7 (30.0) | 16.7 (29.4)
  Cycle 8 (n=33, 22) | 43.4 (31.7) | 15.9 (26.5)
  Cycle 9 (n=33, 18) | 40.4 (29.8) | 14.8 (20.5)
  Cycle 10 (n=29, 14) | 40.2 (32.6) | 9.5 (15.6)
Statistical Analysis 1: Comparison: Sunitinib vs Placebo; Cycle 2 through Cycle 10; Test type: Superiority or Other; p < 0.0001, Repeated Measures Mixed-Effects Model — [p-value comment as in outcome 6, analysis 1]; Mean Difference (Final Values) = 21.3801, 95% CI 2-sided [14.3 to 28.4] — [estimate comment as in outcome 6, analysis 1]

15. Secondary Outcome: EORTC QLQ-C30 - Dyspnea Subscale
Description: as for outcome 6
Time Frame: Day 1 and every 4 weeks thereafter (Day 1 of each 4-week cycle) and at end of treatment/withdrawal
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Sunitinib | Placebo
Number analyzed (Participants) | 73 | 71
scores on a scale
  Cycle 1 (n=67, 66) | 15.9 (21.2) | 19.7 (29.2)
  Cycle 2 (n=69, 66) | 23.2 (26.4) | 22.7 (29.3)
  Cycle 3 (n=60, 56) | 20.6 (24.6) | 20.8 (30.2)
  Cycle 4 (n=55, 43) | 25.5 (26.4) | 22.5 (27.9)
  Cycle 5 (n=48, 41) | 20.8 (27.2) | 16.3 (22.5)
  Cycle 6 (n=42, 30) | 19.0 (23.4) | 15.6 (31.2)
  Cycle 7 (n=38, 28) | 19.3 (24.1) | 19.6 (26.1)
  Cycle 8 (n=34, 22) | 22.5 (28.1) | 21.2 (30.1)
  Cycle 9 (n=32, 18) | 25.0 (25.4) | 18.5 (28.5)
  Cycle 10 (n=29, 14) | 18.4 (26.1) | 16.7 (25.3)
Statistical Analysis 1: Comparison: Sunitinib vs Placebo; Cycle 2 through Cycle 10; Test type: Superiority or Other; p = 0.1339, Repeated Measures Mixed-Effects Model — [p-value comment as in outcome 6, analysis 1]; Mean Difference (Final Values) = 5.2300, 95% CI 2-sided [-1.6 to 12.1] — [estimate comment as in outcome 6, analysis 1]

16. Secondary Outcome: EORTC QLQ-C30 - Fatigue Subscale
Description: as for outcome 6
Time Frame: Day 1 and every 4 weeks thereafter (Day 1 of each 4-week cycle) and at end of treatment/withdrawal
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Sunitinib | Placebo
Number analyzed (Participants) | 73 | 71
scores on a scale
  Cycle 1 (n=67, 66) | 29.4 (23.7) | 34.5 (26.4)
  Cycle 2 (n=69, 67) | 44.3 (24.2) | 40.1 (30.1)
  Cycle 3 (n=60, 56) | 41.2 (23.6) | 42.3 (32.6)
  Cycle 4 (n=55, 43) | 41.0 (26.0) | 37.0 (29.5)
  Cycle 5 (n=48, 41) | 34.7 (23.4) | 36.3 (31.8)
  Cycle 6 (n=42, 31) | 34.9 (25.9) | 42.3 (33.1)
  Cycle 7 (n=38, 28) | 36.5 (24.9) | 34.9 (27.2)
  Cycle 8 (n=34, 22) | 39.9 (28.4) | 43.2 (33.0)
  Cycle 9 (n=33, 18) | 37.4 (22.5) | 37.7 (27.8)
  Cycle 10 (n=29, 14) | 33.7 (23.7) | 43.7 (30.3)
Statistical Analysis 1: Comparison: Sunitinib vs Placebo; Cycle 2 through Cycle 10; Test type: Superiority or Other; p = 0.6138, Repeated Measures Mixed-Effects Model — [p-value comment as in outcome 6, analysis 1]; Mean Difference (Final Values) = 1.7816, 95% CI 2-sided [-5.1 to 8.7] — [estimate comment as in outcome 6, analysis 1]

17. Secondary Outcome: EORTC QLQ-C30 - Financial Difficulties Subscale
Description: as for outcome 6
Time Frame: Day 1 and every 4 weeks thereafter (Day 1 of each 4-week cycle) and at end of treatment/withdrawal
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Sunitinib | Placebo
Number analyzed (Participants) | 73 | 71
scores on a scale
  Cycle 1 (n=67, 66) | 19.9 (32.3) | 15.7 (27.6)
  Cycle 2 (n=68, 65) | 14.2 (26.0) | 14.4 (26.3)
  Cycle 3 (n=59, 56) | 15.8 (25.8) | 16.7 (28.4)
  Cycle 4 (n=55, 43) | 18.2 (27.8) | 12.4 (27.2)
  Cycle 5 (n=48, 40) | 18.1 (28.3) | 13.3 (24.8)
  Cycle 6 (n=42, 30) | 19.0 (29.6) | 11.1 (23.7)
  Cycle 7 (n=38, 28) | 20.2 (33.4) | 10.7 (22.3)
  Cycle 8 (n=34, 22) | 18.6 (32.0) | 13.6 (19.7)
  Cycle 9 (n=33, 18) | 20.2 (26.3) | 14.8 (28.5)
  Cycle 10 (n=29, 14) | 17.2 (29.0) | 14.3 (31.3)
Statistical Analysis 1: Comparison: Sunitinib vs Placebo; Cycle 2 through Cycle 10; Test type: Superiority or Other; p = 0.9367, Repeated Measures Mixed-Effects Model — [p-value comment as in outcome 6, analysis 1]; Mean Difference (Final Values) = 0.2778, 95% CI 2-sided [-6.6 to 7.1] — [estimate comment as in outcome 6, analysis 1]

18. Secondary Outcome: EORTC QLQ-C30 - Insomnia Subscale
Description: as for outcome 6
Time Frame: Day 1 and every 4 weeks thereafter (Day 1 of each 4-week cycle) and at end of treatment/withdrawal
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Sunitinib | Placebo
Number analyzed (Participants) | 73 | 71
scores on a scale
  Cycle 1 (n=67, 66) | 25.4 (29.6) | 26.3 (27.7)
  Cycle 2 (n=69, 67) | 36.7 (35.8) | 27.4 (30.7)
  Cycle 3 (n=59, 56) | 35.6 (30.9) | 24.7 (27.2)
  Cycle 4 (n=55, 43) | 35.2 (33.0) | 22.5 (24.9)
  Cycle 5 (n=48, 41) | 25.0 (26.2) | 24.0 (27.4)
  Cycle 6 (n=42, 30) | 31.0 (32.4) | 28.9 (35.8)
  Cycle 7 (n=38, 28) | 32.9 (35.6) | 23.2 (29.2)
  Cycle 8 (n=34, 22) | 28.4 (34.9) | 28.8 (23.7)
  Cycle 9 (n=33, 18) | 26.3 (32.0) | 29.6 (30.0)
  Cycle 10 (n=29, 14) | 31.0 (34.4) | 23.8 (24.2)
Statistical Analysis 1: Comparison: Sunitinib vs Placebo; Cycle 2 through Cycle 10; Test type: Superiority or Other; p = 0.0372, Repeated Measures Mixed-Effects Model — [p-value comment as in outcome 6, analysis 1]; Mean Difference (Final Values) = 7.7530, 95% CI 2-sided [0.5 to 15] — [estimate comment as in outcome 6, analysis 1]

19. Secondary Outcome: EORTC QLQ-C30 - Nausea and Vomiting Subscale
Description: as for outcome 6
Time Frame: Day 1 and every 4 weeks thereafter (Day 1 of each 4-week cycle) and at end of treatment/withdrawal
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Sunitinib | Placebo
Number analyzed (Participants) | 73 | 71
scores on a scale
  Cycle 1 (n=67, 66) | 6.7 (12.3) | 12.6 (22.1)
  Cycle 2 (n=69, 67) | 13.0 (19.6) | 16.4 (21.8)
  Cycle 3 (n=60, 56) | 15.8 (22.6) | 15.3 (25.4)
  Cycle 4 (n=55, 43) | 15.8 (21.4) | 15.1 (24.1)
  Cycle 5 (n=48, 41) | 15.6 (25.1) | 11.6 (15.9)
  Cycle 6 (n=42, 31) | 11.5 (16.7) | 14.5 (17.6)
  Cycle 7 (n=38, 28) | 13.8 (19.6) | 9.5 (16.0)
  Cycle 8 (n=34, 22) | 11.8 (22.3) | 16.3 (25.0)
  Cycle 9 (n=33, 18) | 9.6 (16.7) | 6.5 (11.6)
  Cycle 10 (n=29, 14) | 8.6 (14.5) | 3.6 (9.6)
Statistical Analysis 1: Comparison: Sunitinib vs Placebo; Cycle 2 through Cycle 10; Test type: Superiority or Other; p = 0.6939, Repeated Measures Mixed-Effects Model — [p-value comment as in outcome 6, analysis 1]; Mean Difference (Final Values) = 1.1463, 95% CI 2-sided [-4.6 to 6.9] — [estimate comment as in outcome 6, analysis 1]

20. Secondary Outcome: EORTC QLQ-C30 - Pain Subscale
Description: as for outcome 6
Time Frame: Day 1 and every 4 weeks thereafter (Day 1 of each 4-week cycle) and at end of treatment/withdrawal
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Sunitinib | Placebo
Number analyzed (Participants) | 73 | 71
scores on a scale
  Cycle 1 (n=67, 66) | 22.9 (24.4) | 22.5 (28.9)
  Cycle 2 (n=69, 67) | 29.5 (27.6) | 28.6 (34.5)
  Cycle 3 (n=60, 56) | 28.1 (27.4) | 28.7 (32.0)
  Cycle 4 (n=55, 43) | 25.5 (27.9) | 24.0 (28.7)
  Cycle 5 (n=48, 41) | 26.7 (25.4) | 28.0 (32.8)
  Cycle 6 (n=42, 31) | 25.0 (25.6) | 31.2 (34.1)
  Cycle 7 (n=38, 28) | 23.9 (26.9) | 23.5 (25.6)
  Cycle 8 (n=34, 22) | 23.0 (26.6) | 28.0 (33.1)
  Cycle 9 (n=33, 18) | 25.3 (24.7) | 22.2 (32.8)
  Cycle 10 (n=29, 14) | 17.2 (15.7) | 26.2 (26.7)
Statistical Analysis 1: Comparison: Sunitinib vs Placebo; Cycle 2 through Cycle 10; Test type: Superiority or Other; p = 0.3711, Repeated Measures Mixed-Effects Model — [p-value comment as in outcome 6, analysis 1]; Mean Difference (Final Values) = -3.5128, 95% CI 2-sided [-11.2 to 4.2] — [estimate comment as in outcome 6, analysis 1]

ADVERSE EVENTS:
Arm/Group | Sunitinib | Placebo
Serious Adverse Events (participants affected / at risk) | 22/83 | 34/82
Other Adverse Events (participants affected / at risk) | 80/83 | 70/82
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sunitinib (N=83) | Placebo (N=82)
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Cardiac failure (Cardiac disorders) | 2 | 0
Ventricular arrhythmia (Cardiac disorders) | 1 | 0
Eye disorder (Eye disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 4
Abdominal pain upper (Gastrointestinal disorders) | 2 | 0
Ascites (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Duodenal ulcer (Gastrointestinal disorders) | 1 | 1
Duodenal ulcer perforation (Gastrointestinal disorders) | 0 | 1
Erosive duodenitis (Gastrointestinal disorders) | 0 | 1
Haematemesis (Gastrointestinal disorders) | 0 | 2
Ileus (Gastrointestinal disorders) | 0 | 1
Mallory-Weiss syndrome (Gastrointestinal disorders) | 1 | 0
Melaena (Gastrointestinal disorders) | 0 | 2
Nausea (Gastrointestinal disorders) | 2 | 1
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1
Varices oesophageal (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 2 | 3
Asthenia (General disorders) | 0 | 1
Disease progression (General disorders) | 3 | 2
Fatigue (General disorders) | 1 | 1
General physical health deterioration (General disorders) | 1 | 2
Hyperthermia (General disorders) | 1 | 0
Inflammation (General disorders) | 0 | 1
Mucosal inflammation (General disorders) | 1 | 0
Multi-organ failure (General disorders) | 0 | 1
Oedema (General disorders) | 0 | 1
Oedema peripheral (General disorders) | 0 | 1
Pyrexia (General disorders) | 1 | 2
Bile duct obstruction (Hepatobiliary disorders) | 1 | 0
Cholangitis (Hepatobiliary disorders) | 0 | 1
Hepatic failure (Hepatobiliary disorders) | 0 | 2
Hepatic function abnormal (Hepatobiliary disorders) | 1 | 0
Hepatic pain (Hepatobiliary disorders) | 1 | 2
Anal abscess (Infections and infestations) | 1 | 0
Catheter related infection (Infections and infestations) | 1 | 0
Liver abscess (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1
Varicella (Infections and infestations) | 1 | 0
Accident (Injury, poisoning and procedural complications) | 0 | 1
Facial bones fracture (Injury, poisoning and procedural complications) | 0 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 1
Joint sprain (Injury, poisoning and procedural complications) | 0 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 | 0
Stent occlusion (Injury, poisoning and procedural complications) | 0 | 1
Therapeutic agent toxicity (Injury, poisoning and procedural complications) | 0 | 1
Traumatic brain injury (Injury, poisoning and procedural complications) | 0 | 1
Haemoglobin decreased (Investigations) | 0 | 1
Lipase increased (Investigations) | 1 | 0
Acidosis (Metabolism and nutrition disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cerebral haematoma (Nervous system disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 1
Convulsion (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 1 | 0
Hepatic encephalopathy (Nervous system disorders) | 1 | 1
Leukoencephalopathy (Nervous system disorders) | 1 | 0
Somnolence (Nervous system disorders) | 0 | 1
Renal failure (Renal and urinary disorders) | 2 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Deep vein thrombosis (Vascular disorders) | 0 | 1
Hypertension (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 0 | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sunitinib (N=83) | Placebo (N=82)
Anaemia (Blood and lymphatic system disorders) | 4 | 8
Leukopenia (Blood and lymphatic system disorders) | 8 | 1
Neutropenia (Blood and lymphatic system disorders) | 23 | 3
Thrombocytopenia (Blood and lymphatic system disorders) | 13 | 4
Hypothyroidism (Endocrine disorders) | 6 | 1
Eyelid oedema (Eye disorders) | 6 | 0
Abdominal pain (Gastrointestinal disorders) | 23 | 23
Abdominal pain upper (Gastrointestinal disorders) | 10 | 6
Aphthous stomatitis (Gastrointestinal disorders) | 5 | 2
Constipation (Gastrointestinal disorders) | 12 | 16
Diarrhoea (Gastrointestinal disorders) | 48 | 32
Dry mouth (Gastrointestinal disorders) | 7 | 5
Dyspepsia (Gastrointestinal disorders) | 12 | 5
Flatulence (Gastrointestinal disorders) | 5 | 2
Gingival bleeding (Gastrointestinal disorders) | 7 | 0
Haemorrhoids (Gastrointestinal disorders) | 5 | 0
Nausea (Gastrointestinal disorders) | 36 | 24
Oral pain (Gastrointestinal disorders) | 5 | 0
Stomatitis (Gastrointestinal disorders) | 18 | 2
Vomiting (Gastrointestinal disorders) | 28 | 24
Asthenia (General disorders) | 28 | 22
Chest pain (General disorders) | 5 | 5
Chills (General disorders) | 8 | 2
Fatigue (General disorders) | 27 | 21
Mucosal inflammation (General disorders) | 13 | 6
Oedema (General disorders) | 5 | 2
Oedema peripheral (General disorders) | 10 | 11
Pyrexia (General disorders) | 9 | 7
Urinary tract infection (Infections and infestations) | 6 | 3
Blood alkaline phosphatase increased (Investigations) | 3 | 6
Weight decreased (Investigations) | 13 | 9
Anorexia (Metabolism and nutrition disorders) | 18 | 17
Decreased appetite (Metabolism and nutrition disorders) | 5 | 4
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2 | 7
Hypoglycaemia (Metabolism and nutrition disorders) | 8 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 5 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 12 | 5
Back pain (Musculoskeletal and connective tissue disorders) | 10 | 14
Muscle spasms (Musculoskeletal and connective tissue disorders) | 5 | 4
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 6 | 8
Pain in extremity (Musculoskeletal and connective tissue disorders) | 8 | 5
Dizziness (Nervous system disorders) | 5 | 5
Dysgeusia (Nervous system disorders) | 17 | 4
Headache (Nervous system disorders) | 15 | 11
Depression (Psychiatric disorders) | 2 | 5
Insomnia (Psychiatric disorders) | 15 | 10
Cough (Respiratory, thoracic and mediastinal disorders) | 7 | 7
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 10 | 12
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 17 | 4
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 6 | 2
Alopecia (Skin and subcutaneous tissue disorders) | 5 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 12 | 9
Erythema (Skin and subcutaneous tissue disorders) | 8 | 4
Hair colour changes (Skin and subcutaneous tissue disorders) | 24 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 3 | 6
Nail disorder (Skin and subcutaneous tissue disorders) | 8 | 1
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 19 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 4 | 9
Rash (Skin and subcutaneous tissue disorders) | 15 | 4
Yellow skin (Skin and subcutaneous tissue disorders) | 6 | 0
Hypertension (Vascular disorders) | 22 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of < 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), < 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.